CLINICAL TRIAL: NCT01163526
Title: Perfusion CT as a Predictor of Treatment Response in Patients With Hepatic Malignancies
Status: Terminated | Type: Observational
Why Stopped: accrual
Sponsor: Stanford University (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry); GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: HEP0031; SU-07092010-6491 (Other: Stanford University)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Neuroendocrine Tumors; Brain (Nervous System) Cancers; Colon/Rectal Cancer; Colon Cancer; Hepatobiliary Cancers; Hepatocellular Carcinoma (Hepatoma); Liver
MeSH Terms: conditions — Neuroendocrine Tumors; Neurologic Manifestations; Neoplasms; Colonic Neoplasms; Carcinoma, Hepatocellular | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- neuroendocrine metastases: 15 patients with neuroendocrine metastases
  Interventions: Procedure: CT perfusion
- colon cancer metastases: 15 patients with colon cancer metastases
  Interventions: Procedure: CT perfusion
- HCC treated with cyberknife radiation and chemotherapy: 15 patients with HCC treated with cyberknife radiation and chemotherapy
  Interventions: Procedure: CT perfusion
- HCC treated with Sirsphere embolization and chemotherapy: 15 patients with HCC treated with Sirsphere embolization and chemotherapy
  Interventions: Procedure: CT perfusion

INTERVENTIONS:
Procedure: CT perfusion

SUMMARY:
A research study of liver perfusion (how blood flows to the liver over time). We hope to learn whether perfusion characteristics of liver masses may be predictive of response to treatment and whether liver perfusion characteristics can be used to follow response to treatment.

ELIGIBILITY:
Inclusion Criteria:3.1.1 Patients with suspected or biopsy-proven liver masses including unresectable hepatocellular carcinoma (HCC), unresectable colon cancer metastases to the liver, and metastatic neuroendocrine tumors to the liver will be eligible for enrollment.

3.1.2 Patients who have undergone prior chemotherapy more than one year prior to the study are eligible for enrollment.

3.1.4 Patients must be 18 years or older. Patients must not be pregnant and, if of child-bearing age, must take precautions not to become pregnant.

3.1.5 No life expectancy restrictions.

3.1.6 ECOG and Karnofsky Performance Status will not be employed.

3.1.7 Patients with renal failure are ineligible for this study (Glomerular filtration rate (GFR) must be > 60)

3.1.8 Ability to understand and willingness to sign a written informed consent document. Exclusion Criteria:3.2.1 Patients who have undergone prior chemoembolization of hepatocellular carcinoma (HCC) are ineligible for enrollment. Patients who have undergone chemotherapy within one year prior to the study are also ineligible for enrollment.

3.2.2 No restrictions regarding use of other investigational agents.

3.2.3 Patients with severe contrast allergy are ineligible.

3.2.4 Patients who are pregnant or are trying to become pregnant are excluded from this study.

3.2.5 Patients who are cancer survivors or Human Immunodeficiency Virus (HIV)-positive will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be 18 years or older. Patients must not be pregnant and, if of child-bearing age, must take precautions not to become pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Predict RECIST response to treatment | at 3 months from CT perfusion parameters before and after treatment

SECONDARY OUTCOMES:
Characterize CT perfusion longitudinally in both responders and nonresponders | 1 yr
Predict disease progression | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States